CLINICAL TRIAL: NCT02097823
Title: A Pilot Study Comparing Olanzapine and Aprepitant for the Prevention of Chemotherapy Induced Nausea and Vomiting in Pediatric Patients Receiving Highly Emetogenic Chemotherapy
Brief Title: Pilot Study of Olanzapine and Aprepitant to Prevent Nausea and Vomiting in Children Receiving Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Holly M. Knoderer, M.D., Indiana University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 1401283326
Record Dates: First submitted 2014-03-21; First posted 2014-03-27 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
Keywords: olanzapine; Nausea and vomiting; aprepitant; pediatrics
MeSH Terms: conditions — Vomiting; Nausea | interventions — Olanzapine; Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant First, Olanzapine Second (Experimental): Will receive aprepitant (weight based dose, see below) in first cycle of chemotherapy and olanzapine (weight based dose, see below) in the second cycle of chemotherapy. All doses will be given starting 30 minutes before chemotherapy on day 1.
  Olanzapine dosing:
  >60kg - 10mg orally daily for 4 doses 40-59.9kg - 5mg orally daily for 4 doses 20-39.9kg - 2.5mg orally daily for 4 doses <20kg - 1.25mg orally daily for 4 doses
  Aprepitant dosing:
  >40kg - 125mg orally on day 1, then 80mg orally daily on days 2,3 35-39.9kg - 80mg orally daily for 3 doses 20-34.9kg - 40mg orally daily for 3 doses <20kg - 1.5-2mg/kg orally daily for 3 doses
  Interventions: Drug: Olanzapine; Drug: Aprepitant
- Olanzapine First, Aprepitant Second (Experimental): Will receive olanzapine (weight based dose, see below) in first cycle of chemotherapy and aprepitant (weight based dose, see below) in the second cycle of chemotherapy. All doses will be given starting 30 minutes before chemotherapy on day 1.
  Olanzapine dosing:
  >60kg - 10mg orally daily for 4 doses 40-59.9kg - 5mg orally daily for 4 doses 20-39.9kg - 2.5mg orally daily for 4 doses <20kg - 1.25mg orally daily for 4 doses
  Aprepitant dosing:
  >40kg - 125mg orally on day 1, then 80mg orally daily on days 2,3 35-39.9kg - 80mg orally daily for 3 doses 20-34.9kg - 40mg orally daily for 3 doses <20kg - 1.5-2mg/kg orally daily for 3 doses
  Interventions: Drug: Olanzapine; Drug: Aprepitant

INTERVENTIONS:
Drug: Olanzapine
  Other Names: zyprexa
Drug: Aprepitant
  Other Names: emend

SUMMARY:
The purpose of this study is to determine the feasibility of a larger trial comparing olanzapine and aprepitant and to obtain preliminary data on the effectiveness of these two medications to treat nausea and vomiting in children receiving chemotherapy. Children receiving 2 cycles of chemotherapy with a high risk of causing nausea and vomiting will receive olanzapine in one cycle and aprepitant in another cycle. Children will be randomized to see which medicine they receive first. The investigators will record the number of extra medications used for nausea, the number of times a child vomits, and the amount of nausea the child feels each day.

DETAILED DESCRIPTION:
This will be a pilot study, designed as a randomized, crossover study comparing olanzapine and aprepitant in pediatric oncology patients receiving highly emetogenic chemotherapy (HEC). The primary objective is to determine the feasibility of recruitment and data collection for conducting a larger trial aimed at comparing olanzapine and aprepitant as antiemetic regimens and establishing efficacy of this regimens for pediatric patients receiving HEC. Secondary objectives are to obtain preliminary data regarding the effectiveness of olanzapine and aprepitant as well as the tolerability of olanzapine in the pediatric oncology population.

Each patient must be planned to undergo at least 2 cycles of the same cycle of HEC. Each patient will be randomized to receive olanzapine or aprepitant in the first cycle of chemotherapy, and then will receive the other agent in a second cycle of chemotherapy. Patients will also receive ondansetron and dexamethasone with each cycle. Patients with CNS tumors will not receive dexamethasone. Response will be measured objectively recording number of emesis and use of breakthrough medications. The medications chosen for breakthrough medications will be at the treating physicians discretion. A complete response will be no episodes of emesis or use of breakthrough medications. A partial response is one or less episodes of emesis and one or less use of breakthrough medications. Nausea will be measured based on parent and patient scales and will be a separate measure, not included in the compete or partial response.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 4 years and less than 21 years
* patient will receive at least two cycles of the same regimen of highly emetogenic chemotherapy
* adequate liver function - defined as total bilirubin less than or equal to 1.5 times the upper limit of normal for age and AST/ALT less than or equal to upper limit of normal for age
* adequate kidney function - defined as creatinine clearance or GFR greater than or equal to 70mL/min/1.73m2 or a serum creatinine based on age/gender as follows: Maximum serum creatinine

  * 2- <6 years: Male & Female 0.8
  * 6- <10 years: Male & Female 1
  * 10- <13 years: Male & Female 1.2
  * 13- <16 years: Male 1.5 Female 1.4
  * >16 years: Male 1.7 Female 1.4

Exclusion Criteria:

* known QTc prolongation or other cardiac arrhythmia
* current treatment with another antipsychotic (for example: risperidone, quetiapine, clozapine)
* prior adverse reaction to either olanzapine or aprepitant
* the planned two cycles of chemotherapy include ifosfamide (a patient may receive ifosfamide as a part of his/her overall treatment plan but not during study cycles)

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Knoderer, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant First, Olanzapine Second: Will receive aprepitant (weight based dose, see below) in first cycle of chemotherapy and olanzapine (weight based dose, see below) in the second cycle of chemotherapy. All doses will be given starting 30 minutes before chemotherapy on day 1.
  Olanzapine dosing:
  >60kg - 10mg orally daily for 4 doses 40-59.9kg - 5mg orally daily for 4 doses 20-39.9kg - 2.5mg orally daily for 4 doses <20kg - 1.25mg orally daily for 4 doses
  Aprepitant dosing:
  >40kg - 125mg orally on day 1, then 80mg orally daily on days 2,3 35-39.9kg - 80mg orally daily for 3 doses 20-34.9kg - 40mg orally daily for 3 doses <20kg - 1.5-2mg/kg orally daily for 3 doses
  Olanzapine
  Aprepitant
- Olanzapine First, Aprepitant Second: Will receive olanzapine (weight based dose, see below) in first cycle of chemotherapy and aprepitant (weight based dose, see below) in the second cycle of chemotherapy. All doses will be given starting 30 minutes before chemotherapy on day 1.
  Olanzapine dosing:
  >60kg - 10mg orally daily for 4 doses 40-59.9kg - 5mg orally daily for 4 doses 20-39.9kg - 2.5mg orally daily for 4 doses <20kg - 1.25mg orally daily for 4 doses
  Aprepitant dosing:
  >40kg - 125mg orally on day 1, then 80mg orally daily on days 2,3 35-39.9kg - 80mg orally daily for 3 doses 20-34.9kg - 40mg orally daily for 3 doses <20kg - 1.5-2mg/kg orally daily for 3 doses
  Olanzapine
  Aprepitant
Period: Overall Study
Arm/Group | Aprepitant First, Olanzapine Second | Olanzapine First, Aprepitant Second
Started | 11 | 4
Completed | 10 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant First, Olanzapine Second | Olanzapine First, Aprepitant Second | Total
Number analyzed (Participants) | 11 | 4 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 3 | 14
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 10.5 [5 to 14] | 14 [13 to 18] | 11.8 [5 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 6 | 2 | 8
Diagnosis [Number; unit: participants]
  Ewings | 2 | 2 | 4
  Osteosarcoma | 3 | 1 | 4
  Neuroblastoma | 2 | 0 | 2
  Hodgkins | 2 | 0 | 2
  Germ Cell Tumor | 1 | 0 | 1
  Histiocytic Sarcoma | 0 | 1 | 1
  Medulloblastoma | 1 | 0 | 1
Chemotherapy Regimen [Number; unit: participants]
  Vincristine/Cyclophosphamide/Doxorubicin | 2 | 2 | 4
  Cisplatin/Doxorubicin | 2 | 1 | 3
  High Dose Methotrexate | 1 | 0 | 1
  Cisplatin/Etoposide | 2 | 0 | 2
  BEACOPP | 1 | 0 | 1
  ABVE-PC | 1 | 0 | 1
  Cisplatin/Bleomycin/Etoposide | 1 | 0 | 1
  CHOP | 0 | 1 | 1
  Cisplatin/Vincristine | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment and Data Collection.
Description: Primary objective of this study is to determine the feasibility of recruitment and data collection for conducting a larger trial. Recruitment and data collection will be feasible if at least 20 subjects can be recruited in 1 year and there is a 90% form completion rate.
Time Frame: Approximately 1 year after study opens, at the conclusion of data collection. Participants will be followed during 2 cycles of chemotherapy, an expected average of 6 weeks. Data will be collected over 5 days during each cycle.
Measure: Number; unit: percentage of completed forms
Units Other Than Participants: Administered forms
Groups:
- All Participants: Both intervention arms included
Arm/Group | All Participants
Number analyzed (Participants) | 14
Number analyzed (Administered forms) | 27
percentage of completed forms | 70.4

2. Secondary Outcome: Complete Response in Overall Phase
Description: This will measure what percentage of patients have a complete response (no emesis or use of breakthrough medications) in the overall phase (0-120 hours).
Time Frame: Participants will be followed during 2 cycles of chemotherapy, an expected average of 6 weeks. Data will be collected over 5 days during each cycle.
Measure: Number; unit: percentage of participants with CR
Groups:
- Aprepitant: Cycles where patients received aprepitant along with dexamethasone and ondansetron (regardless of whether cycle 1 or cycle 2)
- Olanzapine: Cycles where patients received olanzapine along with dexamethasone and ondansetron (regardless of whether cycle 1 or cycle 2)
Arm/Group | Aprepitant | Olanzapine
Number analyzed (Participants) | 13 | 14
percentage of participants with CR | 23.1 | 28.6

3. Secondary Outcome: Complete Response in Acute Phase
Description: This will measure what percentage of patients have a complete response (no emesis or use of breakthrough medications) in the acute phase (0-24 hours).
Time Frame: as for outcome 2
Measure: Number; unit: percentage of participants with CR
Arm/Group | Aprepitant | Olanzapine
Number analyzed (Participants) | 13 | 14
percentage of participants with CR | 76.9 | 78.6

4. Secondary Outcome: Complete Response in Delayed Phase
Description: This will measure what percentage of patients have a complete response (no emesis or use of breakthrough medications) in the delayed phase (25-120 hours).
Time Frame: as for outcome 2
Measure: Number; unit: percentage of participants with CR
Arm/Group | Aprepitant | Olanzapine
Number analyzed (Participants) | 13 | 14
percentage of participants with CR | 23.1 | 28.6

5. Secondary Outcome: Good Control of Nausea
Description: Good control of nausea will be ratings <25 on visual analog scale by parents and <2 on baxter retching faces scale by patients. Will look at the proportions of patients with good control of nausea.
  The visual analog scale ranged from 0-100, with 0 being no nausea and 100 being very very severe nausea. The Baxter retching faces scale ranged from 0-10 using only even numbers (0,2,4,6,8,10) and each number has a corresponding face depicting someone experiencing varying levels of nausea, with 0 being no nausea and 10 being a picture of face vomiting.
Time Frame: as for outcome 2
Population: could only analyze cycles where subjects had returned completed forms
Measure: Number; unit: percentage of participant w/good control
Arm/Group | Aprepitant | Olanzapine
Number analyzed (Participants) | 11 | 8
percentage of participant w/good control
  Visual Analog Scale/Parents | 54.5 | 50
  BARF scale/Patients | 54.5 | 50

6. Other Pre Specified Outcome: Number of Participants With Adverse Events.
Description: Olanzapine will be considered tolerable if less than 10% of patients experience a grade III or IV adverse event attributable to olanzapine.
Time Frame: Ongoing, throughout the study. Will be fully evaluated in approximately 1 year, at the conclusion of data collection. Each patient will be followed during 2 cycles of chemotherapy, an expected average of 6 weeks.
Measure: Number; unit: participants
Arm/Group | Aprepitant | Olanzapine
Number analyzed (Participants) | 13 | 14
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Aprepitant | Olanzapine
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant (N=15) | Olanzapine (N=15)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2) — Grade I agitation

LIMITATIONS AND CAVEATS:
This trial was a pilot study, limited by numbers of participants. Given the small numbers, during randomization (with 50/50 chance each subject randomized to group A or B) a disproportionate number of patients were randomized to group A.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes